CLINICAL TRIAL: NCT00040365
Title: Amifostine as a Rectal Protector During External Beam Radiotherapy for Prostate Cancer: A Phase II Study
Brief Title: Amifostine to Protect the Rectum During External Beam Radiotherapy for Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Kevin A. Camphausen, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 020215; 02-C-0215; NCT00045253 (obsolete NCT alias)
Record Dates: First submitted 2002-06-25; First posted 2002-06-26 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Radiation Therapy; Rectal Toxicity; Amifostine; Radioprotector
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Amifostine; Radiotherapy; Radiation; X-Ray Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amifostine (Experimental): 1000 mg for the first 18 patients. 2000 mg for the last 12 patients. The syringe of amifostine will be connected to a rectal enema bottle for administration. Administered slowly over 30-60 seconds with the patient in recumbent position 30-45 minutes prior to each radiation treatment (33-39 doses).
  Interventions: Drug: Amifostine trihydrate; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Amifostine trihydrate — 1000 mg for the first 18 patients. 2000 mg for the last 12 patients. The syringe of amifostine will be connected to a rectal enema bottle for administration. Administered slowly over 30-60 seconds with the patient in recumbent position 30-45 minutes prior to each radiation treatment (33-39 doses).
  Other Names: Ethyol
Radiation: Radiation therapy — The treatment will be delivered in at least two phases. The first field reduction will occur after 46Gy and the second field reduction will occur after 70Gy.
  Other Names: radiotherapy; irradiation; x-ray therapy

SUMMARY:
This study will evaluate the safety and effectiveness of a drug called amifostine in reducing the bowel side effects of radiation treatment for prostate cancer. Amifostine is a 'radioprotector' medicine that to protects normal tissue from radiation damage. This study will determine whether placing amifostine in the rectum during radiation treatment for prostate cancer can decrease common side effects of treatment, including diarrhea, painful bowel movements, bleeding, and gas.

Patients 18 years of age or older with prostate cancer may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, bone scan if a recent one is not available, and possibly computed tomography (CT) and magnetic resonance imaging (MRI) scans of the pelvis. They will also have a liquid retention test, in which they are given an enema of 4 tablespoons of salt water that they must retain for 20 minutes.

Participants will receive standard radiation therapy for prostate cancer-5 consecutive days for 8 weeks-in the National Institutes of Health (NIH) Radiation Oncology Clinic. Amifostine will be placed in the rectum by a mini-enema before each radiation treatment so that it covers the lining of the rectum. To determine the side effects of the treatment, patients will undergo a proctoscopic examination before beginning radiation therapy, two times during therapy, and at each follow-up visit for 5 years after treatment ends. This examination involves inserting a proctoscope (a thin flexible tube with a light at the end) into the rectum and taking pictures.

Patients will be followed in the clinic at visits scheduled 1, 3, 6, 12, 18, 24, 36, 48, and 60 months after treatment for a physical examination and routine blood tests, proctoscopic examination, and review of bowel symptoms.

DETAILED DESCRIPTION:
Normal tissue tolerance of the rectum limits the dose of radiation that can be delivered to the prostate for curative treatment of prostate cancer. Amifostine is a radioprotector, an agent that reduces tissue damage incurred by ionizing radiation. It has been well studied in humans and is approved for intravenous use. Rectal administration results in a preferential accumulation of Amifostine in the rectal mucosa, and neither free parent compound nor free active metabolite have been detected in systemic circulation. This trial proposes to observe the rate of early and late bowel toxicity in a group of patients with prostate cancer receiving standard high dose, 3D conformal external beam radiotherapy and concurrent intra-rectal applications of Amifostine. Primary measures of rectal toxicity (RTOG radiation morbidity scoring) will also be compared with self-assessment measures of quality of life, and rectal radiation dose as assessed by dose-volume histograms.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pathologically confirmed adenocarcinoma of the prostate gland.

Age greater than or equal to 18 years.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed (this does not include routine laboratory tests or imaging studies required to establish eligibility).

EXCLUSION CRITERIA:

Other active malignancy (except for non-melanoma skin cancer).

Patient with a prior history of pelvic or prostate radiotherapy.

Patients with chronic inflammatory bowel disease.

Patients with distant metastatic disease.

Cognitively impaired patients who cannot give informed consent.

Human Immunodeficiency Virus (HIV) positivity.

Other medical conditions deemed by the principal investigator (PI) or associates to make the patient ineligible for high dose radiotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-06; Primary Completion 2010-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Greenlee RT, Hill-Harmon MB, Murray T, Thun M. Cancer statistics, 2001. CA Cancer J Clin. 2001 Jan-Feb;51(1):15-36. doi: 10.3322/canjclin.51.1.15. PMID 11577478
- [Background] Fuks Z, Leibel SA, Wallner KE, Begg CB, Fair WR, Anderson LL, Hilaris BS, Whitmore WF. The effect of local control on metastatic dissemination in carcinoma of the prostate: long-term results in patients treated with 125I implantation. Int J Radiat Oncol Biol Phys. 1991 Aug;21(3):537-47. doi: 10.1016/0360-3016(91)90668-t. PMID 1869452
- [Background] Pollack A, Smith LG, von Eschenbach AC. External beam radiotherapy dose response characteristics of 1127 men with prostate cancer treated in the PSA era. Int J Radiat Oncol Biol Phys. 2000 Sep 1;48(2):507-12. doi: 10.1016/s0360-3016(00)00620-9. PMID 10974469
- [Result] Simone NL, Menard C, Soule BP, Albert PS, Guion P, Smith S, Godette D, Crouse NS, Sciuto LC, Cooley-Zgela T, Camphausen K, Coleman CN, Singh AK. Intrarectal amifostine during external beam radiation therapy for prostate cancer produces significant improvements in Quality of Life measured by EPIC score. Int J Radiat Oncol Biol Phys. 2008 Jan 1;70(1):90-5. doi: 10.1016/j.ijrobp.2007.05.057. Epub 2007 Sep 12. PMID 17855015
- [Result] Simone, NL; Soule, BP; Ménard, C; Albert, P; Guion, P; Smith, S; Godette, D; Coleman, CN; Singh, AK. Assessing Rectal Toxicity in a Pilot Study using Intrarectal Amifostine and Concurrent Radiation. 42nd annual meeting of the American society of clinical oncology, Atlanta, GA, June 2006.
- [Result] Menard C, Camphausen K, Muanza T, Sears-Crouse N, Smith S, Ben-Josef E, Coleman CN. Clinical trial of endorectal amifostine for radioprotection in patients with prostate cancer: rationale and early results. Semin Oncol. 2003 Dec;30(6 Suppl 18):63-7. doi: 10.1053/j.seminoncol.2003.11.016. PMID 14727242
- [Result] Singh AK, Menard C, Guion P, Simone NL, Smith S, Crouse NS, Godette DJ, Cooley-Zgela T, Sciuto LC, Coleman J, Pinto P, Albert PS, Camphausen K, Coleman CN. Intrarectal amifostine suspension may protect against acute proctitis during radiation therapy for prostate cancer: a pilot study. Int J Radiat Oncol Biol Phys. 2006 Jul 15;65(4):1008-13. doi: 10.1016/j.ijrobp.2006.02.030. Epub 2006 May 26. PMID 16730138
- [Result] Simone NL, Ménard C, Singh AK, Guion P, Smith S, Crouse NS, Godette D, Cooley-Zgela T, Sciuto LC, Coleman J, Pinto, P, Albert PS, Camphausen K, Coleman CN. Intrarectal amifostine suspension may protect against acute proctitis during radiation therapy for prostate cancer: oral presentation at 91st scientific assembly and annual meeting of the radiological society of North America, Chicago, IL, 2005.
- [Result] Muanza TM, Albert PS, Smith S, Godette D, Crouse NS, Cooley-Zgela T, Sciuto L, Camphausen K, Coleman CN, Menard C. Comparing measures of acute bowel toxicity in patients with prostate cancer treated with external beam radiation therapy. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1316-21. doi: 10.1016/j.ijrobp.2004.12.083. PMID 16029787
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0215.html
- See also: Medline Plus — http://www.nlm.nih.gov/medlineplus/
- See also: Drug Information — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial accrued 30 participants.
Period: Overall Study
Arm/Group | Amifostine
Started | 30
Completed Follow Up Phase | 19
Completed | 19
Not Completed | 11
Not completed — Death | 1
Not completed — Progressive disease | 7
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Amifostine
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 65.63 (7.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 2
  Black | 2
  White | 23
  Hispanic | 3
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Good Toxicity Outcome Who Experienced an Acute Rectal Toxicity and Received Topical Administrations of Amifostine in Conjunction With High Dose, 3D Conformal Radiotherapy for Prostate Cancer.
Description: A good toxicity outcome is defined as having less than grade 2 on both weeks 5 and 7 of treatment. The Radiation Therapy Oncology Group (RTOG) Acute radiation morbidity scoring scheme and the Rectal Mucosal Toxicity response criteria will be used to assess rectal toxicity. The RTOG measures the rectal toxicities. The physician assigns a grade based on symptoms reported by the patient. For details about the RTOG (method and scoring of radiation morbidity, etc.) see http://www.rtog.org/ResearchAssociates/AdverseEventReporting/AcuteRadiationMorbidityScoringCriteria.aspx
Time Frame: RTOG Acute was used on week 5 and 7
Population: Number of participants 29 versus 30 = One patient was taken off study due to tumor progression prior to the follow up period.
Measure: Number; unit: Percentage of Participants
Arm/Group | Amifostine
Number analyzed (Participants) | 29
Percentage of Participants | 20.69

2. Secondary Outcome: Percentage of Participants With a Good Toxicity Outcome Who Experienced Late Rectal Toxicity and Received Topical Administrations of Amifostine in Conjunction With High Dose, 3D Conformal Radiotherapy for Prostate Cancer.
Description: A good toxicity outcome is defined as having less than grade 2 on both weeks 5 and 7 of treatment. Week 5, 7 were during treatment measuring acute toxicity. The Radiation Therapy Oncology Group (RTOG) Acute radiation morbidity scoring scheme and the Rectal Mucosal Toxicity response criteria will be used to assess rectal toxicity. The RTOG measures the rectal toxicities. The physician assigns a grade based on symptoms reported by the patient. For details about the RTOG see http://www.rtog.org/ResearchAssociates/AdverseEventReporting/AcuteRadiationMorbidityScoringCriteria.aspx.
Time Frame: The late rectal toxicity has been assessed at 1, 3, 6, 12, 18, 24, 36, and 60 months after the completion of treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Amifostine
Number analyzed (Participants) | 6
Percentage of Participants | 83.33

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 3 years
Measure: Number; unit: Participants
Arm/Group | Amifostine
Number analyzed (Participants) | 30
Participants | 30

4. Secondary Outcome: Expanded Prostate Cancer Index Composite (EPIC) Bowel Assessment Over Time (Late Follow-up 18 Months)
Description: The EPIC bowel assessment is a 26 item short form evaluation that assess patient function and bother after prostate treatment. The Expanded Prostate Cancer Index Composite is a self assessment questionnaire designed to measure quality of life in patients with prostate cancer. The questionnaire is scored on a scale of 0-100 with higher scores correlated with higher function and quality of life. For this study, the Bowel Domain was analyzed alongside the RTOG acute and late gastrointestinal morbidity scores. For details re: EPIC, see http://www.med.umich.edu/urology/research/EPIC/EPIC-2.2002.pdf
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amifostine
Number analyzed (Participants) | 30
scores on a scale | 0.6 (0.1)

5. Secondary Outcome: Measures of Quality of Life (QOL)-(Late Follow-up 18 Months)
Description: Radiation toxicity consists of the Radiation Therapy Oncology Group(RTOG)acute(within 90 days of treatment)and RTOG late(>90days after treatment). This scoring system assigns a toxicity grade (0-4) based on symptoms with 0 being the best outcome. The Expanded Prostate Cancer Index Composite(EPIC) questionnaire consists of 50 quality of life items divided into 4 domains, urinary, bowel, sexual and hormonal. Each independent domain renders a scoring of 0-100 with 100 being the best score. The EPIC and RTOG scores were correlated not combined.
Time Frame: Baseline, week 5, 7 , and months 1, 3, 6, 12, and 18
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Amifostine
Number analyzed (Participants) | 30
scores on a scale
  Baseline bowel function | 91.13 [71.43 to 100]
  Baseline bowel bother | 92.86 [67.86 to 100]
  Week 5 bowel function | 71.43 [39.29 to 96.43]
  Week 5 bowel bother | 67.33 [28.57 to 100]
  Week 5 RTOG | 1.06 [0 to 2]
  Week 7 bowel function | 69.76 [32.14 to 100]
  Week 7 bowel bother | 66.38 [21.43 to 96.43]
  Week 7 RTOG | 1.00 [0 to 2]
  1 month bowel function | 84.09 [42.86 to 100]
  1 month bowel bother | 78.08 [32.14 to 96.43]
  1 month RTOG | 0.59 [0 to 1]
  3 month bowel function | 79.08 [46.43 to 100]
  3 month bowel bother | 82.78 [17.86 to 100]
  3 month RTOG | 0.54 [0 to 2]
  6 month bowel function | 85.46 [50 to 100]
  6 month bowel bother | 81.86 [50 to 100]
  6 month RTOG | 0.39 [0 to 1]
  12 month bowel function | 83.92 [39.29 to 100]
  12 month bowel bother | 77.65 [10.71 to 100]
  12 month RTOG | 0.50 [0 to 2]
  18 month bowel function | 83.55 [50 to 100]
  18 month bowel bother | 76.28 [14.29 to 100]
  18 month RTOG | 0.64 [0 to 2]

6. Secondary Outcome: Number of Participants Who Had Proctoscopic Examinations
Description: Proctoscopic scoring of mucosal change was performed according to a descriptive scale, described by Wachter et al, which assigns grades of mucosal congestion, telangiectasia, ulcerations, stricture, and necrosis.
Time Frame: 3 years
Measure: Number; unit: Participants
Arm/Group | Amifostine
Number analyzed (Participants) | 30
Participants | 30

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Amifostine
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amifostine (N=30)
Proctitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amifostine (N=30)
abdominal pain/cramping (Reproductive system and breast disorders) | 4 (5) — Common Toxicity Criteria (CTC) v2.0 Adverse Event (AE)
allergic reaction/hypersensitivity (Immune system disorders) | 1 (1) — CTCv2.0 AE
alopecia (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) — CTCv2.0 AE
bladder (Renal and urinary disorders) | 1 (1) — CTCv2.0 AE
cardiac-ischemia/infarction (Cardiac disorders) | 1 (1) — CTCv2.0 AE
chest pain (Nervous system disorders) | 1 (1) — CTCv2.0 AE
chills (General disorders) | 1 (1) — CTCv2.0 AE
CN. VI (Nervous system disorders) | 1 (1) — CTCv2.0 AE
Constipation (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) — CTCv2.0 AE
diarrhea (Gastrointestinal disorders) | 25 (42) — CTCv2.0 AE
Dry mouth (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
dry skin (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) — CTCv2.0 AE
dysuria (Renal and urinary disorders) | 16 (24) — CTCv2.0 AE
erectile dysfunction (Reproductive system and breast disorders) | 3 (3) — CTCv2.0 AE
erectile impotence (Reproductive system and breast disorders) | 18 (24) — CTCv2.0 AE
erythema (Skin and subcutaneous tissue disorders) | 3 (3) — CTCv2.0 AE
fatigue (General disorders) | 27 (48) — CTCv2.0 AE
flatulence (Gastrointestinal disorders) | 9 (9) — CTCv2.0 AE
Genitourinary (Renal and urinary disorders) | 1 (1) — CTCv2.0 AE
headache (Nervous system disorders) | 1 (1) — CTCv2.0 AE
hematochezia (Blood and lymphatic system disorders) | 6 (7) — CTCv2.0 AE
hematuria (Renal and urinary disorders) | 4 (5) — CTCv2.0 AE
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
Hot Flashes (Endocrine disorders) | 1 (1) — CTCv2.0 AE
hot flashes/flushes (Endocrine disorders) | 5 (10) — CTCv2.0 AE
hypotension (Vascular disorders) | 1 (1) — CTCv2.0 AE
incontinence (Renal and urinary disorders) | 23 (34) — CTCv2.0 AE
injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
insomnia (Psychiatric disorders) | 2 (2) — CTCv2.0 AE
Knee (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
libido (Reproductive system and breast disorders) | 6 (6) — CTCv2.0 AE
mood alteration- depression (Nervous system disorders) | 22 (34) — CTCv2.0 AE
mucositis (Gastrointestinal disorders) | 20 (29) — CTCv2.0 AE
mucous membrane (Gastrointestinal disorders) | 19 (28) — CTCv2.0 AE
nausea (Gastrointestinal disorders) | 3 (4) — CTCv2.0 AE
neck/shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
neuropathy-sensory (Nervous system disorders) | 3 (4) — CTCv2.0 AE
orgasmic dysfunction (Reproductive system and breast disorders) | 1 (1) — CTCv2.0 AE
other-weak stream (ibuprofen) (Renal and urinary disorders) | 20 (32) — CTCv2.0 AE
other- back (d/t bulge disc (L1-L2P) (Musculoskeletal and connective tissue disorders) | 2 (2) — CTCv2.0 AE
other-body hair loss (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
other-breast tenderness (Reproductive system and breast disorders) | 3 (3) — CTCv2.0 AE
other-burning (burning with urination; burning in penis; Cipro) (Renal and urinary disorders) | 1 (3) — CTCv2.0 AE
other-edema (mucosal edema; redness) (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
other-ejaculate (Cipro) (Reproductive system and breast disorders) | 3 (3) — CTCv2.0 AE
other-knee injury (orthopedic evaluation) (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
other-L arm (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
other-L side (Nervous system disorders) | 1 (1) — CTCv2.0 AE
other-local swelling (r/t IL-2 injection) (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
other-low back (d/t osteophytes (MRI); Celebrex; Advil) (Musculoskeletal and connective tissue disorders) | 1 (1) — CTCv2.0 AE
other-mucositis (erythema) (Gastrointestinal disorders) | 2 (3) — CTCv2.0 AE
other-pressure (incr pressure urinary stream) (Renal and urinary disorders) | 1 (1) — CTCv2.0 AE
other-rectal spasm (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
other-tenesmus (Gastrointestinal disorders) | 2 (2) — CTCv2.0 AE
other-tubular adenoma (colonoscopy/bx 12/19/05) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — CTCv2.0 AE
Pain: Headaches (Nervous system disorders) | 1 (1) — CTCv2.0 AE
palpitations (Cardiac disorders) | 1 (1) — CTCv2.0 AE
proctitis (Gastrointestinal disorders) | 29 (89) — CTCv2.0 AE
pruritis (Skin and subcutaneous tissue disorders) | 8 (9) — CTCv2.0 AE
radiation dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — CTCv2.0 AE
sm/ lg bowel (Gastrointestinal disorders) | 28 (89) — CTCv2.0 AE
syncope (Nervous system disorders) | 1 (1) — CTCv2.0 AE
taste disturbance (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
thrombosis/embolism (Vascular disorders) | 1 (1) — CTCv2.0 AE
Tremor-arms (Nervous system disorders) | 1 (1) — CTCv2.0 AE
urinary frequency/urgency (Renal and urinary disorders) | 27 (57) — CTCv2.0 AE
urinary retention (Renal and urinary disorders) | 21 (36) — CTCv2.0 AE
vomiting (Gastrointestinal disorders) | 1 (1) — CTCv2.0 AE
weight gain (General disorders) | 13 (20) — CTCv2.0 AE
weight loss (General disorders) | 11 (11) — CTCv2.0 AE
Bladder (Renal and urinary disorders) | 1 (1) — Radiation Therapy Oncology Group (RTOG) Adverse Event (AE)
Mucous membrane (Skin and subcutaneous tissue disorders) | 19 (28) — RTOG AE
Small/large bowel (Gastrointestinal disorders) | 28 (89) — RTOG AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No